CLINICAL TRIAL: NCT00965224
Title: Therapeutic Efficacy of Wilms Tumor Gene (WT1) MRNA-electroporated Autologous Dendritic Cell Vaccination in Patients with Myeloid Malignancies and Multiple Myeloma: a Phase II Trial
Brief Title: Efficacy of Dendritic Cell Therapy for Myeloid Leukemia and Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zwi Berneman (Other)
Responsible Party: Sponsor-Investigator, Zwi Berneman, Professor Dr. Zwi Berneman, University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCRG 09-003
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Acute Myeloid Leukemia; Chronic Myeloid Leukemia; Multiple Myeloma
Keywords: AML (acute myeloid leukemia); CML (chronic myeloid leukemia); MM (multiple myeloma)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- standard therapy + vaccination (Experimental)
  Interventions: Biological: dendritic cell vaccination (active specific immunotherapy)

INTERVENTIONS:
Biological: dendritic cell vaccination (active specific immunotherapy)

SUMMARY:
Dendritic cell therapy is a promising strategy for adjuvant cancer therapy in the setting of minimal residual disease (MRD) to fight off cancer relapse and/or progression. The investigators already performed a phase I safety study in leukemia patients that were in complete remission demonstrating the absence of side effects and feasibility of the therapy. Here, the investigators want to extend on this strategy by studying the clinical efficacy of autologous DC vaccination in patients with acute and chronic myeloid leukemia and myeloma patients. Effects of DC therapy on the immune reactivity towards leukemia cells as well as clinical parameters such molecular MRD monitoring, time to relapse (TTR), progression-free survival (PFS) and overall survival(OS) will be studied in vaccinated and non-vaccinated (control) patients. Patients will be vaccinated using their own dendritic cells electroporated with mRNA coding for the full-length Wilms' tumor antigen WT1.

ELIGIBILITY:
Inclusion Criteria:

* Acute Myeloid Leukemia (AML): all FAB subtypes except M3. Extent of disease:

  * clinical remission after at least one course of polychemotherapy
  * high risk of relapse due to age (> 60 years) or poor risk cytogenetic/molecular markers or hyperleukocytosis at presentation or previous relapse
* Chronic myeloid leukemia (CML): patients in chronic phase under therapy with tyrosinase kinase inhibitors who have sub-optimal response or failure and who are not eligible for hematopoietic stem cell transplantation.
* Multiple Myeloma (MM): symptomatic with active disease, independent of earlier and/or concomitant treatment:

  * Presence of serum/urine M protein (> 3 g/dl)
  * Bone marrow plasmacytosis (>10-30%)
  * Anemia, renal failure, hypercalcemia, and/or lytic bone lesions
* Overexpression of WT1 RNA in peripheral blood and or bone marrow as assessed by quantitative RT-PCR at the time of presentation.For CML: residual molecular disease as demonstrated by BCR-ABL RT-PCR
* Prior treatments: Patients must have received at least one prior antileukemic chemotherapeutic regimen and must be more than 1 month past the last treatment.
* Age: ≥ 18 years
* Performance status: WHO PS grade 0-1 (Appendix B)
* Objectively assessable parameters of life expectancy: more than 3 months
* Prior and concomitant associated diseases allowed with the exception of underlying autoimmune disease and positive serology for HIV/HBV/HCV
* No concomitant use of immunosuppressive drugs
* adequate renal and liver function, i.e. creatinin and bilirubin = 1.2 times the upper limit of normal
* absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Women of child-bearing potential should use adequate contraception prior to study entry and for the duration of study participation

Exclusion Criteria:

* Subjects with concurrent additional malignancy (with exception of non-melanoma skin cancers and carcinoma in situ of the cervix)
* Subjects who are pregnant
* Subjects who have sensitivity to drugs that provide local anesthesia
* Subjects needing corticosteroids 1 mg/kg during vaccination; corticosteroids are allowed as part of their treatment when taken ≥ 30 days before the start of vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of WT1 mRNA-transfected DC vaccination | Upon completion of blood sample collection (before start of the vaccination at week 0 and 8 weeks after start of the vaccination) and skin biopsy collection (8 weeks after start of the vaccination) for all included patients
Induction/maintenance of molecular remission as evidenced by molecular MRD monitoring of WT1 (AML, CML and MM) and BCR/ABL RNA (CML) copies in peripheral blood | Upon follow-up completion for all included patients, i.e. until 24 months after the last vaccination

SECONDARY OUTCOMES:
Time to relapse (TTR) | Upon follow-up completion for all included patients, i.e. until 24 months after the last vaccination
progression-free survival | Upon follow-up completion for all included patients, i.e. until 24 months after the last vaccination
overall survival (OS) | Upon follow-up completion for all included patients, i.e. until 24 months after the last vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

REFERENCES:
- [Background] Van Driessche A, Van de Velde AL, Nijs G, Braeckman T, Stein B, De Vries JM, Berneman ZN, Van Tendeloo VF. Clinical-grade manufacturing of autologous mature mRNA-electroporated dendritic cells and safety testing in acute myeloid leukemia patients in a phase I dose-escalation clinical trial. Cytotherapy. 2009;11(5):653-68. doi: 10.1080/14653240902960411. PMID 19530029
- [Background] Smits EL, Berneman ZN, Van Tendeloo VF. Immunotherapy of acute myeloid leukemia: current approaches. Oncologist. 2009 Mar;14(3):240-52. doi: 10.1634/theoncologist.2008-0165. Epub 2009 Mar 16. PMID 19289488
- [Background] Van Driessche A, Gao L, Stauss HJ, Ponsaerts P, Van Bockstaele DR, Berneman ZN, Van Tendeloo VF. Antigen-specific cellular immunotherapy of leukemia. Leukemia. 2005 Nov;19(11):1863-71. doi: 10.1038/sj.leu.2403930. PMID 16121214
- [Background] Smits EL, Anguille S, Cools N, Berneman ZN, Van Tendeloo VF. Dendritic cell-based cancer gene therapy. Hum Gene Ther. 2009 Oct;20(10):1106-18. doi: 10.1089/hum.2009.145. PMID 19656053
- [Derived] Anguille S, Van de Velde AL, Smits EL, Van Tendeloo VF, Juliusson G, Cools N, Nijs G, Stein B, Lion E, Van Driessche A, Vandenbosch I, Verlinden A, Gadisseur AP, Schroyens WA, Muylle L, Vermeulen K, Maes MB, Deiteren K, Malfait R, Gostick E, Lammens M, Couttenye MM, Jorens P, Goossens H, Price DA, Ladell K, Oka Y, Fujiki F, Oji Y, Sugiyama H, Berneman ZN. Dendritic cell vaccination as postremission treatment to prevent or delay relapse in acute myeloid leukemia. Blood. 2017 Oct 12;130(15):1713-1721. doi: 10.1182/blood-2017-04-780155. Epub 2017 Aug 22. PMID 28830889